CLINICAL TRIAL: NCT03970122
Title: A First-In-Human, Phase 1, Placebo-Controlled Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of GFB-887, a TRPC5 Channel Inhibitor, in Healthy Subjects
Brief Title: FIH Ph 1 Study of TRPC5 Channel Inhibitor GFB-887 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Goldfinch Bio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: GFB-887-101; 8391348 (Other: Covance)
Record Dates: First submitted 2019-05-24; First posted 2019-05-31 (Actual); Last update posted 2020-06-02 (Actual); Status verified 2020-06

CONDITIONS: Healthy Volunteers
Keywords: Glomerulosclerosis; proteinuria; nephrotic syndrome; nephrosis; focal segmental glomerulosclerosis; kidney diseases; urologic diseases; glomerulonephritis; nephritis; diabetic kidney disease; diabetic nephropathies; endocrine system diseases; diabetes complications
MeSH Terms: conditions — Proteinuria; Nephrotic Syndrome; Nephrosis; Glomerulosclerosis, Focal Segmental; Kidney Diseases; Urologic Diseases; Glomerulonephritis; Nephritis; Diabetic Nephropathies; Endocrine System Diseases; Diabetes Complications

STUDY DESIGN:
Intervention Model Description: Dose escalation, parallel assignment
Who Masked: Participant, Investigator
Masking Description: Blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- GFB-887 SAD active (Experimental): GFB-887 single dose active
  Interventions: Drug: GFB-887
- GFB-887 SAD placebo (Placebo Comparator): GFB-887 single dose placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GFB-887 — IMP
  Arms: GFB-887 SAD active
Drug: Placebo — Matching
  Arms: GFB-887 SAD placebo

SUMMARY:
The study will comprise primarily a single-ascending dose (SAD) escalation component.

DETAILED DESCRIPTION:
Double-blind, randomized, placebo-controlled, single-dose, sequential-group design in up to 7 cohorts of healthy participants.

ELIGIBILITY:
Healthy Participant Cohorts - Key Inclusion Criteria:

1. Males or females, of any race, between 18 and 55 years of age, inclusive, at Screening.
2. Body mass index between 18.0 and 32.0 kg/m^2, inclusive, at Screening.
3. Systolic blood pressure of between 90 and 140 mmHg, diastolic blood pressure between 60 and 90 mmHg, and heart rate between 40 and 100 bpm at Screening.
4. Female participants will be post-menopausal or surgically sterile (as confirmed by medical history).
5. Male participants will agree to use contraception while on study drug and for at least 90 days after the final follow-up visit.
6. Able to comprehend and willing to sign an informed consent form (ICF) and to abide by the study restrictions.
7. Participants must be in good health.

Healthy Participant Cohorts - Key Exclusion Criteria:

1. Females of childbearing potential.
2. Significant history or clinically significant manifestation of any metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, respiratory, endocrine, or psychiatric disorder, as determined by the Investigator (or designee).
3. History of alcoholism or drug/chemical abuse within 2 years prior to (first) Check-in.
4. Use of tobacco or nicotine-containing products within 60 days prior to (first) dosing, or positive cotinine at Screening or Check-in.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Males, females of non-childbearing potential
Enrollment: 70 (Actual)
Dates: Start 2019-05-29 (Actual); Primary Completion 2020-03-04 (Actual); Study Completion 2020-04-04 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of AEs | Approximately 5.5 weeks
  Safety and tolerability
Incidence of clinically significant changes in laboratory parameters, 12 lead ECG parameters, vital signs measurements, spirometry, and physical examinations | Approximately 5.5 weeks
  Safety and tolerability
Plasma PK parameters: Cmax | Approximately 5.5 weeks
  PK
Plasma PK parameters: Tmax | Approximately 5.5 weeks
  PK
Plasma PK parameters: AUC | Approximately 5.5 weeks
  PK
Urine PK parameters: Ae | Approximately 5.5 weeks
  PK
Urine PK parameters: Fe | Approximately 5.5 weeks
  PK
Urine PK parameters: CLR | Approximately 5.5 weeks
  PK

CONTACTS AND LOCATIONS:
Overall Officials: Jeanelle Kam, MD, Principal Investigator — Covance Clinical Research Unit
Locations (1):
- Covance Clinical Research Unit Inc., Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No